CLINICAL TRIAL: NCT02767895
Title: A Pilot Trial of Prehabilitation Among Patients Undergoing PAD Revascularization
Brief Title: Prehabilitation for PAD Revascularization Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment and change in available study resources
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth A. Jackson, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00113096
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Peripheral Vascular Disease; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): Participants will be referred to the Michigan Surgical & Health Optimization Program in the month leading up to their surgery. Individuals are encouraged to increase their physical activity, practice stress reduction, and other behaviors associated with good health
  Interventions: Behavioral: Prehabilitation
- Usual Care (No Intervention): Participants will follow the pre-operative instructions provided by their surgical team.

INTERVENTIONS:
Behavioral: Prehabilitation — Participants will receive an informational DVD, a pedometer, an incentive spirometer and access to the program website to help promote healthful behaviors and improved well-being in the days leading up to surgery.
  Other Names: MSHOP - Michigan Surgical & Health Optimization Program
  Arms: Prehabilitation

SUMMARY:
Patients undergoing elective revascularization of their peripheral artery disease will be randomized to a prehabilitation program or usual care prior to their scheduled procedure.

DETAILED DESCRIPTION:
Patients undergoing elective revascularization for their peripheral artery disease will be randomized to a "prehabilitation" program prior to their surgery or to usual care. The prehabilitation program is self-directed program designed to improve health and quality of life prior to surgery. The program is currently offered to general surgery patients; this study will examine the feasibility and acceptability of such a program in a different patient population.

ELIGIBILITY:
Inclusion Criteria:

* Documented lower extremity PAD
* Ability to walk at least 1 block
* Sedentary
* Medical clearance from the surgical team
* Competent to provide consent

Exclusion Criteria:

* Life expectancy < 6 months
* Co-morbidities which limit walking to a severe degree
* Signs of critical limb ischemia
* Recent or current enrollment in a formal exercise program
* Recent cardiovascular events including stroke, TIA, severe valve disease, etc.
* Current substance abuse
* Psychiatric disorder which limits ability to participate in study procedures
* Non-English speaking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of Study as Indicated by Number of Participants | 1 day
  The feasibility of the study will be assessed by analyzing the recruitment of subjects to the study and the compliance of recruited subjects to the protocol. Feasibility will be defined as able to screening, approaching, and enrolling 25 eligible patients to the pilot study.
Acceptability of Study as Indicated by Percentage of Participation | 8 months
  The willingness of patients to enroll and complete the basic study procedures. Acceptability will be defined as low drop out-rates (<15%), completion of quality of life surveys, and >85% usage of the pedometers.

SECONDARY OUTCOMES:
Increased Physical Activity Characteristics | 8 months
  Increased physical activity characteristics will be assessed through the Godin Leisure Time and International Physical Activity Questionnaire, and questionnaires on barriers to and self-efficacy of exercise.
Health-related Quality of Life | 8 months
  Health-related quality of life and physical activity characteristics will be measured during the pre, peri, and post-operative period. This will be done through PROMIS surveys, which assess physical function, fatigue, depression, anxiety, and ability to participate in and satisfaction with social roles/activities.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jackson, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No